CLINICAL TRIAL: NCT01869764
Title: A Randomized, Placebo-Controlled Phase II Clinical Trial of Omega-3 PUFA Dietary Supplementation in Patients With Stage I-III Breast Carcinoma
Brief Title: Omega-3 Fatty Acid in Treating Patients With Stage I-III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00023419; NCI-2013-00963 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 98113 (Other: NCI)
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ; Male Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms, Male; Breast Neoplasms | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (omega-3 fatty acid) (Experimental): Patients receive omega-3 fatty acid PO daily for 7-14 days.
  Interventions: Drug: omega-3 fatty acid; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO daily for 7-14 days.
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: omega-3 fatty acid — Given PO
  Other Names: fish oil; n-3 fatty acid; O3FA
  Arms: Arm I (omega-3 fatty acid)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II clinical trial studies how well omega-3 fatty acid works in treating patients with stage I-III breast cancer. Studying samples of tissue and blood in the laboratory from breast cancer patients receiving omega-3 fatty acid may help doctors learn more about the effects of omega-3 fatty acid on tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if omega-3 dietary supplementation (omega-3 fatty acid) results in higher polyunsaturated fatty acids (PUFA) levels in surgical specimens of normal and malignant breast tissue in women who took omega 3 tablets in comparison to those who took placebo.

II. To determine if omega-3 dietary supplementation results in higher PUFA levels in plasma and red blood cells in women who took omega 3 tablets in comparison to those who took placebo.

III. To determine if omega-3 dietary supplementation affects the metabolites of omega-3 and omega-6 PUFA in surgical specimens of malignant and normal breast tissue in comparison to controls.

IV. To determine if women who take omega-3 dietary supplementation have less proliferation and greater apoptosis in malignant breast tissue in comparison to women who take placebo.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive omega-3 fatty acid orally (PO) daily for 7-14 days.

ARM II: Patients receive placebo PO daily for 7-14 days.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage I to III breast cancer and carcinoma in situ (including lobular carcinoma in situ [LCIS] and ductal carcinoma in situ [DCIS])
* Breast surgery (lumpectomy or mastectomy) is planned for at least 7 days from the day of enrollment
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved written informed consent document
* Tumor measures at least 1 centimeter on imaging or physical exam

Exclusion Criteria:

* Any patient with surgery scheduled < 7days after biopsy
* Patients who are unable to refrain from the use of any NSAID or full-dose acetylsalicylic acid (ASA)-containing NSAID while taking study drug
* Patients who will receive neoadjuvant chemotherapy are not eligible
* Patients who are currently taking omega-3 fatty acids, as they are unable to be randomized to placebo
* Patients who have previously taken omega-3 fatty acid within 1 month prior to study enrollment
* Patients with an allergy or known hypersensitivity to fish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Levine, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
Started | 28 | 29
Completed | 28 | 27
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo) | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (14.0) | 59.9 (9.5) | 58.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 23 | 23 | 46
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: PUFA Levels in Normal and Metastatic Breast Tissue
Description: Analysis of variance (ANOVA) will be used to assess the effect of omega-3 dietary supplementation on PUFA levels separately in normal and malignant breast tissue. Analysis of covariance (ANCOVA) will be used to assess the omega-3 effect in plasma and red blood cells (RBC), where the baseline levels of the PUFAs will be included as covariates. PUFA Levels analyzed were 18:2 n-6, 18:3 n-3, 20:2 n-6, 20:4 n-6, 20:3 n-3, 20:5 n-3, 22:6 n-3
Time Frame: At time of surgery
Population: All samples measurements were not available for all participants to be analyzed.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 22 | 19
ug/ml
  Normal breast tissue 18:2 n-6 | 60.986 (40.392) | 72.762 (50.742)
  Normal breast tissue 18:3 n-3 | 3.232 (2.289) | 3.505 (2.041)
  Normal breast tissue 20:2 n-6 | 1.104 (0.96) | 1.008 (0.724)
  Normal breast tissue 20:4 n-6 | 2.221 (1.349) | 2.342 (1.445)
  Normal breast tissue 20:3 n-3 | 0.049 (0.107) | 0.038 (0.085)
  Normal breast tissue 20:5 n-3 | 0.027 (0.128) | 0.034 (0.147)
  Normal breast tissue 22:6 n-3 | 0.095 (0.443) | 0.061 (0.264)
  Normal breast tissue n-3 | 3.402 (2.572) | 3.64 (2.24)
  Normal breast tissue n-6 | 3.421 (2.085) | 3.413 (1.962)
  Normal breast tissue n3/n-6 ratio: number analyzed (Participants) | 21 | 19
  Normal breast tissue n3/n-6 ratio | 0.948 (0.468) | 1.102 (0.438)
  Malignant breast tissue 18:2 n-6 | 44.137 (44.544) | 33.735 (31.548)
  Malignant breast 18:3 n-3 | 1.943 (2.162) | 1.356 (1.465)
  Malignant breast 20:2 n-6 | 0.889 (0.886) | 0.601 (0.657)
  Malignant breast 20:4 n-6 | 3.208 (1.948) | 2.248 (1.744)
  Malignant breast 20:3 n-3 | 0.034 (0.087) | 0 (0)
  Malignant breast 20:5 n-3 | 0.2 (0.665) | 0 (0)
  Malignant breast 22:6 n-3 | 0 (0) | 0 (0)
  Malignant breast n-3 | 2.178 (2.41) | 1.357 (1.466)
  Malignant breast n-6 | 48.233 (46.105) | 36.586 (32.856)
  Malignant breast n-3/n-6 ratio | 0.029 (0.031) | 0.032 (0.016)
  Differences in PUFA level 18:2 n-6 | -16.85 (51.043) | -39.027 (38.697)
  Differences in PUFA level 18:3 n-3 | -1.289 (2.784) | -2.149 (1.935)
  Differences in PUFA level 20:2 n-6 | -0.215 (0.866) | -0.407 (0.514)
  Differences in PUFA level 20:4 n-6 | 0.986 (1.595) | -0.094 (1.589)
  Differences in PUFA level 20:3 n-3 | -0.015 (0.105) | -0.038 (0.085)
  Differences in PUFA level 20:5 n-3 | 0.173 (0.545) | -0.034 (0.147)
  Differences in PUFA level 22:6 n-3 | -0.095 (0.443) | -0.061 (0.264)
  Difference in PUFA level n-3 | -1.224 (2.794) | -2.282 (2.127)
  Difference in PUFA level in n-6 | 44.812 (45.463) | 33.173 (31.836)
  Difference in n-3/n-6 ratio: number analyzed (Participants) | 21 | 19
  Difference in n-3/n-6 ratio | -0.92 (0.45) | -1.07 (0.438)

2. Primary Outcome: PUFA Levels in Plasma Pre and Post Surgery
Description: as for outcome 1
Time Frame: Pre and post surgery
Population: All samples measurements were not available for all participants to be analyzed.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 24 | 19
ug/ml
  Plasma pre-surgery 18:2 n-6 | 1514890 (370945) | 1539300 (370726)
  Plasma pre-surgery 18:3 n-3 | 37501 (25256) | 33119 (19368)
  Plasma pre-surgery 20:2 n-6 | 7039 (6213) | 6031 (5612)
  Plasma pre-surgery 20:4 n-6 | 210238 (77734) | 210006 (83260)
  Plasma pre-surgery 20:3 n-3 | 0 (0) | 0 (0)
  Plasma pre-surgery 20:5 n-3 | 38539 (30967) | 50206 (41170)
  Plasma pre-surgery 22:6 n-3 | 132887 (68619) | 111798 (79889)
  Plasma pre-surgery n-3 | 208297 (105288) | 195123 (106007)
  Plasma pre-surgery n-6 | 1732167 (373713) | 1755338 (397402)
  Plasma pre-surgery n3/n-6 ratio | 0.121 (0.058) | 0.11 (0.049)
  Plasma post-surgery 18:2 n-6: number analyzed (Participants) | 23 | 18
  Plasma post-surgery 18:2 n-6 | 1504732 (497732) | 1507750 (419001.5)
  Plasma post-surgery 18:3 n-3: number analyzed (Participants) | 23 | 18
  Plasma post-surgery 18:3 n-3 | 37472 (18521) | 34202.78 (15615)
  Plasma post-surgery 20:2 n-6: number analyzed (Participants) | 23 | 18
  Plasma post-surgery 20:2 n-6 | 5980 (5351) | 6851.409 (5479.023)
  Plasma post-surgery 20:4 n-6: number analyzed (Participants) | 23 | 18
  Plasma post-surgery 20:4 n-6 | 168100 (63105) | 204127.2 (85101.33)
  Plasma post-surgery 20:3 n-3: number analyzed (Participants) | 23 | 18
  Plasma post-surgery 20:3 n-3 | 0 (0) | 0 (0)
  Plasma post-surgery 20:5 n-3: number analyzed (Participants) | 23 | 18
  Plasma post-surgery 20:5 n-3 | 74521 (48954) | 52643.85 (32019.8)
  Plasma post-surgery 22:6 n-3: number analyzed (Participants) | 23 | 18
  Plasma post-surgery 22:6 n-3 | 153607 (83888) | 133832.8 (74361.31)
  Plasma post-surgery n-3: number analyzed (Participants) | 23 | 18
  Plasma post-surgery n-3 | 265600 (134862) | 220679.4 (108607.5)
  Plasma post-surgery n-6: number analyzed (Participants) | 23 | 18
  Plasma post-surgery n-6 | 1678812 (538264) | 1718729 (448393)
  Plasma post-surgery n-3/n-6 ratio: number analyzed (Participants) | 23 | 18
  Plasma post-surgery n-3/n-6 ratio | 0.16 (0.067) | 0.126 (0.049)
  Differences in PUFA level 18:2 n-6: number analyzed (Participants) | 23 | 18
  Differences in PUFA level 18:2 n-6 | -23266 (602402) | -34877 (365683)
  Differences in PUFA level 18:3 n-3: number analyzed (Participants) | 23 | 18
  Differences in PUFA level 18:3 n-3 | -554 (36051) | 1583 (20838)
  Differences in PUFA level 20:2 n-6: number analyzed (Participants) | 23 | 18
  Differences in PUFA level 20:2 n-6 | -824 (7018) | 485 (5683)
  Differences in PUFA level 20:4 n-6: number analyzed (Participants) | 23 | 18
  Differences in PUFA level 20:4 n-6 | -37844 (87910) | -8045 (69960)
  Differences in PUFA level 20:3 n-3: number analyzed (Participants) | 23 | 18
  Differences in PUFA level 20:3 n-3 | 0 (0) | 0 (0)
  Differences in PUFA level 20:5 n-3: number analyzed (Participants) | 23 | 18
  Differences in PUFA level 20:5 n-3 | 35551 (38628) | 2291 (25409)
  Differences in PUFA level 22:6 n-3: number analyzed (Participants) | 23 | 18
  Differences in PUFA level 22:6 n-3 | 21487 (68743) | 19001 (72461)
  Difference in PUFA level n-3: number analyzed (Participants) | 23 | 18
  Difference in PUFA level n-3 | 56484 (119807) | 22874 (83246)
  Difference in PUFA level in n-6: number analyzed (Participants) | 23 | 18
  Difference in PUFA level in n-6 | -61935 (653885) | -42437 (414325)
  Difference in n-3/n-6 ratio: number analyzed (Participants) | 23 | 18
  Difference in n-3/n-6 ratio | 0.039 (0.056) | 0.015 (0.041)

3. Primary Outcome: PUFA Levels in Red Blood Cells Pre and Post Surgery
Description: as for outcome 1
Time Frame: Pre and post surgery
Population: All samples measurements were not available for all participants to be analyzed.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 20 | 18
ug/ml
  Red blood cells pre-surgery 18:2 n-6 | 351125 (130630) | 387455 (119089)
  Red blood cells pre-surgery 18:3 n-3 | 3430 (4505) | 3211 (4026)
  Red blood cells pre-surgery 20:2 n-6 | 2826 (3515) | 4014 (4183)
  Red blood cells pre-surgeryy 20:4 n-6 | 132624 (68691) | 144208 (71426)
  Red blood cells pre-surgery 20:3 n-3 | 0 (0) | 0 (0)
  Red blood cells pre-surgery 20:5 n-3 | 9723 (13112) | 11005 (14840)
  Red blood cells pre-surgery 22:6 n-3 | 79934 (77518) | 90668 (74168)
  Red blood cells pre-surgery n-3 | 0 (0) | 0 (0)
  Red blood cells pre-surgery n-6 | 0 (0) | 0 (0)
  Red blood cells pre-surgery n3/n-6 ratio | 0 (0) | 0 (0)
  Red blood cells post-surgery 18:2 n-6: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery 18:2 n-6 | 391882 (183779) | 373679 (103361)
  Red blood cells post-surgery 18:3 n-3: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery 18:3 n-3 | 5320 (4709) | 2103 (5007)
  Red blood cells post-surgery 20:2 n-6: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery 20:2 n-6 | 3922 (3941) | 1842 (3315)
  Red blood cells post-surgery 20:4 n-6: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery 20:4 n-6 | 149267 (70598) | 116868 (73523)
  Red blood cells post-surgery 20:3 n-3: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery 20:3 n-3 | 0 (0) | 0 (0)
  Red blood cells post-surgery 20:5 n-3: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery 20:5 n-3 | 25301 (29112) | 9818 (20929)
  Red blood cells post-surgery 22:6 n-3: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery 22:6 n-3 | 110198 (90038) | 64117 (96118)
  Red blood cells post-surgery n-3: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery n-3 | 0 (0) | 0 (0)
  Red blood cells post-surgery n-6: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery n-6 | 0 (0) | 0 (0)
  Red blood cells post-surgery n-3/n-6 ratio: number analyzed (Participants) | 19 | 18
  Red blood cells post-surgery n-3/n-6 ratio | 0 (0) | 0 (0)
  Differences in PUFA level 18:2 n-6: number analyzed (Participants) | 19 | 18
  Differences in PUFA level 18:2 n-6 | 35856 (213680) | -13776 (134998)
  Differences in PUFA level 18:3 n-3: number analyzed (Participants) | 19 | 18
  Differences in PUFA level 18:3 n-3 | 1709 (4746) | -1109 (5750)
  Differences in PUFA level 20:2 n-6: number analyzed (Participants) | 19 | 18
  Differences in PUFA level 20:2 n-6 | 948 (3481) | -2172 (5204)
  Differences in PUFA level 20:4 n-6: number analyzed (Participants) | 19 | 18
  Differences in PUFA level 20:4 n-6 | 23282 (94096) | -27340 (117792)
  Differences in PUFA level 20:3 n-3: number analyzed (Participants) | 19 | 18
  Differences in PUFA level 20:3 n-3 | 0 (0) | 0 (0)
  Differences in PUFA level 20:5 n-3: number analyzed (Participants) | 19 | 18
  Differences in PUFA level 20:5 n-3 | 15066 (29266) | -1187 (28583)
  Differences in PUFA level 22:6 n-3: number analyzed (Participants) | 19 | 18
  Differences in PUFA level 22:6 n-3 | 42086 (101629) | -26551 (128776)
  Difference in PUFA level n-3: number analyzed (Participants) | 19 | 18
  Difference in PUFA level n-3 | 0 (0) | 0 (0)
  Difference in PUFA level in n-6: number analyzed (Participants) | 19 | 18
  Difference in PUFA level in n-6 | 0 (0) | 0 (0)
  Difference in n-3/n-6 ratio: number analyzed (Participants) | 19 | 18
  Difference in n-3/n-6 ratio | 0 (0) | 0 (0)

4. Secondary Outcome: Metabolites of Omega-3 and Omega-6 PUFA in Malignant and Normal Breast Tissue
Description: ANOVA will be used to assess the effect in normal and malignant breast tissue. Metabolites tested: PGE2, PGD2, 20-HETE, 5-HEPE, 13-HODE, 9-HODE, 15-HETE, 12-HETE, 5-HETE.
Time Frame: At time of surgery
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 23 | 19
ug/ml
  Normal breast tissue PGE2 | 9.14 (24.59) | 1.12 (4.5)
  Normal breast tissue PGD2 | 4.47 (16.17) | 2.27 (9.32)
  Normal breast tissue 20HETE | 1.43 (6.87) | 4.24 (18.47)
  Normal breast tissue 13HODE | 4881.23 (11979.79) | 2308.05 (4654.22)
  Normal breast tissue 9HODE | 729.38 (1789.68) | 335.48 (643.24)
  Normal breast tissue 15HETE | 13.99 (28.41) | 28.12 (79.73)
  Normal breast tissue 12HETE | 12.05 (11.37) | 7.87 (8.86)
  Normal breast tissue 5HETE | 4.75 (4.47) | 84.07 (354.6)
  Malignant breast tissue PGE2 | 328.12 (884.633) | 81.15 (181.54)
  Malignant breast tissue PGD2 | 335.88 (894.77) | 92.01 (184.18)
  Malignant breast tissue 20HETE | 11.52 (44.5) | 11.49 (48.06)
  Malignant breast tissue 13HODE | 4584.87 (10465.02) | 2343.46 (4379.73)
  Malignant breast tissue 9HODE | 694.78 (1611.17) | 350.07 (655.21)
  Malignant breast tissue 15HETE | 91.11 (199.85) | 95.85 (190.12)
  Malignant breast tissue 12HETE | 79.17 (233.57) | 14.52 (15.02)
  Malignant breast tissue 5HETE | 11.7 (21.91) | 5.74 (7.74)
  Difference in PGE2 | 319 (868.1) | 80 (182.1)
  Difference in PGD2 | 331.4 (896.4) | 89.7 (185.6)
  Difference in 20HETE | 10.1 (45.4) | 7.3 (52.5)
  Difference in 13HODE | -296.4 (4812.1) | 35.4 (4412.3)
  Difference in 9HODE | -34.6 (761.9) | 14.6 (673.4)
  Difference in 15HETE | 77.1 (191.4) | 67.7 (210.4)
  Difference in 12HETE | 67.1 (229.4) | 6.7 (15.5)
  Difference in 5HETE | 7 (19.6) | -78.3 (355.4)

5. Secondary Outcome: Number of Days to Establish Difference in Proliferation in Malignant Breast Tissue
Description: ANOVA will be used to assess the effect of the supplementation in malignant breast tissue with less proliferation in malignant breast tissue in comparison to women who took the placebo.
Time Frame: At time of surgery
Measure: Mean (Standard Deviation); unit: Days on treatment
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 27 | 25
Days on treatment | 23.7 (16.6) | 24.2 (23.9)
Statistical Analysis 1: Comparison: Arm I (Omega-3 Fatty Acid) vs Arm II (Placebo); Test type: Other; p = 0.93, ANOVA

6. Secondary Outcome: Number of Days to Establish Increased Apoptosis in Malignant Breast Tissue
Description: ANOVA will be used to assess the effect of the supplementation in malignant breast tissue with greater apoptosis in malignant breast tissue in comparison to women who took the placebo.
Time Frame: At time of surgery
Measure: Mean (Standard Deviation); unit: Days on treatment
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 27 | 25
Days on treatment | 2.6 (2.2) | 3.2 (2.4)
Statistical Analysis 1: Comparison: Arm I (Omega-3 Fatty Acid) vs Arm II (Placebo); Test type: Other; p = 0.29, ANOVA

ADVERSE EVENTS:
Time Frame: 14-21 days after surgery
Arm/Group | Arm I (Omega-3 Fatty Acid) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 2/28 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Omega-3 Fatty Acid) (N=28) | Arm II (Placebo) (N=27)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT01869764/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT01869764/ICF_001.pdf